CLINICAL TRIAL: NCT06016036
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study of SAL-0951 Tablets in the Treatment of Renal Anemia in Non-dialysis Chronic Kidney Disease
Brief Title: SAL-0951 Tablets in the Treatment of Renal Anemia in Non-dialysis Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL0951A301
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-08

CONDITIONS: Renal Anemia in Non-dialysis Chronic Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAL-0951 (Experimental)
  Interventions: Drug: SAL-0951
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAL-0951 — SAL-0951：
  1. initial phase：4mg QD for 8 weeks
  2. subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: SAL-0951 group
  Arms: SAL-0951
Drug: Placebo — SAL-0951 placebo：
  1. initial phase：4mg QD for 8 weeks
  2. subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: Placebo phase
  Arms: Placebo

SUMMARY:
This study is a phase 3 randomized, double-blind, placebo-controlled clinical study to evaluate the efficacy and safety of SAL-0951 in CKD-anemia patients in Non-dialysis, comprising 8 weeks of double-blind treatment period followed by an open-label treatment period, making up a total of 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old men and women;
2. 40-100 kg weight;
3. The glomerular filtration rate value calculated by CKD-EPI formula is <60 mL/min/1.73 m^2 (stage 3, 4 or 5 of KDOQI chronic kidney disease) in non-dialyzed subjects with confirmed anemia of chronic kidney disease;
4. Ferritin > 100 g/L and TSAT > 20%;
5. No treatment with ESA was received at least 8 weeks before randomization, and the central laboratory hemoglobin value for the last two screening period (at least 6 days interval) >=80 g/L and <=105 g/L, and the change of absolute value of the two visits <=10g/L;
6. The investigators determined that dialysis or alternative kidney transplantation was not required throughout the trial;
7. Volunteer to participate in the trial and have an informed consent form signed.

Exclusion Criteria:

1. Blood pressure control was poor after regular drug therapy for more than 4 weeks before screening, SBP > 160mmHg or DBP > 100mmHg during screening;
2. Patients with severe complications of hepatobiliary system (AST or ALT > 2.5 ULN, TBiL > 1.5 ULN);
3. Acute kidney injury occurred 12 weeks before screening;
4. NYHA class III - IV heart failure or unstable angina;
5. Acute myocardial infarction, transient ischemic attack, cerebral infarction or pulmonary embolism, deep venous thrombosis occurred 6 months before randomization;
6. Patients requiring ophthalmologic treatment for diabetic eye disease, diabetic macular edema, or age-related macular degeneration, or patients with hypertrophic choroid or retinopathy;
7. Blood transfusion or red blood cell infusion within 3 months before screening;
8. Subjects received protein anabolic hormone, testosterone heptanoate, or methadone within 3 month before screening
9. Severe hyperparathyroidism (iPTH>=500pg/mL);
10. Patients with HIV, HCV or Treponema pallidum antibody positive, or HBsAg positive with HBV DNA>=1000 U/mL;
11. Severe active infection (active tuberculosis, fungal infection, etc.), systemic blood disease (myelodysplastic syndrome, aplastic anemia), or hemolytic anemia, or hemorrhagic anemia;
12. A history of malignancy, exceptions: tumors determined to be cured or in remission for 5 years, skin basal cell or squamous cell carcinomas that have been radically resected, or carcinomas in situ of any site;
13. Chronic inflammatory disease other than glomerulonephritis that may affect red blood cell production, such as systemic lupus erythematosus, rheumatoid arthritis, celiac disease, etc.;
14. A history of severe allergy to medications (e.g. anaphylactic shock) or allergy to other HIF-PH inhibitors;
15. A history of drug or alcohol abuse in the past two years;
16. Participated in clinical trials of any other drug or medical device within 3 months before screening, or plan to participate in any other clinical trials of drug or medical device during the trial;
17. SAL-0951 products or other HIF-PH inhibitors were used before screening;
18. Female during pregnancy or lactation;
19. From the time the informed consent form was sighed to the end of the study, woman of childbearing age who does not agree to use effective contraception, or man whose sexual partner is a woman of childbearing age (Effective methods of contraception include transdermal patches, oral drugs, implantable or injectable contraceptives, abstinence or birth control);
20. Medical conditions that the investigators believe may pose a safety risk to subjects, or confuse efficacy or safety evaluations, or interfere with subject participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Difference in mean Hb concentration levels from baseline at weeks 7-9 | Baseline and week 7-9
  Change From Baseline in mean Hb concentration levels at week 7-9

SECONDARY OUTCOMES:
double-blind phase：The cumulative percentage of subjects who achieved Hb response at any time from treatment to week 9 | Baseline to week 9
  Change From Baseline in cumulative percentage of subjects who achieved Hb response at any time at week 9
Double-blind phase：Proportion of subjects with average Hb level ≥100 g/L at week 7-9 | Week 7-9
Double-blind phase：Proportion of average Hb concentration ≥100g/L and ≤120g/L in week 9 | Week 9
Double-blind phase：By week 9, the cumulative proportion of subjects whose Hb increased by ≥10 g/L and whose Hb reached ≥100g/L | Week 9
Double-blind phase：By week 9, the cumulative proportion of Hb > 130 g/L | Week 9
Double-blind phase：Proportion of subjects receiving intravenous iron at week 9 | Week 9

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No